CLINICAL TRIAL: NCT05866172
Title: A Randomized Controlled Study of Hepatic Arterial Infusion Chemotherapy of FOLFOX With or Without Zoledronic Acid for the Prevention of Bone Metastases in Advanced Hepatocellular Carcinoma Staged at BCLC C
Brief Title: HAIC Combined Withzoledronic Acid for the Prevention of Bone Metastases in Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-069
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; zoledronic Acid; hepatic arterial infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC with zoledronic Acid (Experimental)
  Interventions: Procedure: HAIC; Drug: Zoledronic acid
- HAIC without zoledronic Acid (Active Comparator)
  Interventions: Procedure: HAIC

INTERVENTIONS:
Procedure: HAIC — hepatic arterial infusion of oxaliplatin, LV and 5-fu (20h)
Drug: Zoledronic acid — Zoledronic acid 4mg iv.drip
  Arms: HAIC with zoledronic Acid

SUMMARY:
Zoledronic acid was initially used for bone metastases in various malignancies. However, it is unknown whether hepatic arterial infusion chemotherapy combined with zoledronic acid can improve overall survival of unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Unresectable HCC. For BCLC C HCC, sorafenib/lenvatinib or PD-1/L1 antibody was allowed.
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 8.5 g/dL
* Total bilirubin ≤ 30mmol/L
* Serum albumin ≥ 30 g/L
* ASL and AST ≤ 5 x upper limit of normal
* Serum creatinine ≤ 1.5 x upper limit of normal
* INR ≤ 1.5 or PT/APTT within normal limits
* Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China